CLINICAL TRIAL: NCT03899662
Title: A Neurophysiological Investigation of the Effectiveness of Web-based Exergaming Platform of Cognitive and Physical Training in Schizophrenic Patients
Brief Title: Neurophysiological Evaluation of Schizophrenia Patients After Cognitive and Physical Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Panos Bamidis, Associate Professor, Aristotle University Of Thessaloniki
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: SCH15973
Record Dates: First submitted 2019-03-29; First posted 2019-04-02 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Schizophrenia
Keywords: Electroencephalography; Cognitive training; Physical training; Resting state networks
MeSH Terms: conditions — Schizophrenia | interventions — Cognitive Training; Physical Conditioning, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive and Physical Training (Experimental): 24 sessions (8 weeks, 3 times per week) of computer based 45 minute cognitive and 45 minute physical training.
  Interventions: Other: Cognitive Training; Other: Physical Training

INTERVENTIONS:
Other: Cognitive Training — Cognitive training included memory, attention, velocity, intelligence
Other: Physical Training — Physical training included aerobic, strength, flexibility and balance.

SUMMARY:
Neurophysilogical, neuropsychological evaluation and cognitive and physical training

DETAILED DESCRIPTION:
24 sessions (8 weeks, 3 times per week) of cognitive and physical training via computer. Each session consisted of 45 minutes of cognitive traing (BrainHQ platform https://www.brainhq.com/) and 45 minutes of physical training (FitForAll platform https://www.fitforall.gr/play/app/). Cognitive training included memory, attention, velocity, intelligence etc. Physical training included aerobic, strength flexibility and other excercises. All evaluations were performed 1-14 before the initiation of the interventions and 1-14 after their completion. Neurophysiological evaluation consisted of EEG with the use of 128 electrode-machine and the protocol included 5 minuted of eyes closed and 5 minutes of eyes open. Neuropsychological evaluation included Trail Making Test (A & B), Verbal Fluency, Stroop test, Wechsler Memory - Cubes (visuospatial), MoCA, FAB (Screening for frontal damage) and Eyes Test (Theory of Mind). Also, the physical condition evaluation included 6-Minute Walking Distance (6MWD), ΒΜΙ, HandGrip Strength Test, Short Physical Performance Battery Protocol.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of schizophrenia disorder according to ICD10 criteria
* clinically stable patients (no recent change in psychotropic medication except benzodiazepines)
* sufficient acculturation and fluency in Greek language
* assent of the attending physician for participation in the study

Exclusion Criteria:

* co-morbidity with neurological disorders (e.g.epilepsy) or head injury
* a pathological or other somatic disorder that contraindicate physical exercise
* alcoholism and substance abuse within the previous 3 months (except caffeine and tobacco)
* abstainance from intervention for more than 12 days
* cognitive decline
* treated with Benzodiazepine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Alterations in functional connectivity properties and on the organization of resting state networks | 3 months
  Alterations in functional connectivity properties and on the organization of resting state networks quantified through graph theory tools. These measures would be measured through high-density electroencephalographic (EEG) evaluation and reconstruction of cortical activity.

SECONDARY OUTCOMES:
Physical fitness | 2 months
  Estimated through 6-Minute Walking Distance (6MWD)
Physical fitness | 2 months
  Estimated through ΒΜΙ
Physical fitness | 2 months
  Estimated through HandGrip Strength Test
Physical fitness | 2 months
  Estimated through Short Physical Performance Battery Protocol
Memory | 2 months
  Estimated through Wechsler Memory - Cubes (visuospatial) test
Executive function | 2 months
  Estimated through FAB (Frontalassesment test)
Depressive syndromes | 2 months
  Estimated through Had's test
Theory of mind | 2 months
  Estimated through Eye's test
Verbal fluency | 2 months
  Estimated through Verbal Fluency test
Visual attention and task switching | 2 months
  Estimated through Trail Making A & B test
Reaction time | 2 months
  Estimated through Stroop test
Generic cogntive impairment | 2 months
  Estimated through Montreal Cognitive Assessment (MoCA) test

CONTACTS AND LOCATIONS:
Overall Officials: Panagiotis Bamidis, PhD, Principal Investigator — Associate Professor
Locations (1):
- Laboratory of Medical Physics, AUTH, Thessaloniki, Greece

REFERENCES:
- [Background] Hemsley DR. The development of a cognitive model of schizophrenia: placing it in context. Neurosci Biobehav Rev. 2005;29(6):977-88. doi: 10.1016/j.neubiorev.2004.12.008. PMID 15964074
- [Background] Tagliazucchi E, von Wegner F, Morzelewski A, Borisov S, Jahnke K, Laufs H. Corrigendum to "Automatic sleep staging using fMRI functional connectivity data" [Neuroimage 63/1 (2012) 63-72]. Neuroimage. 2013 Nov 1;81:506. doi: 10.1016/j.neuroimage.2013.05.048. Epub 2013 May 23. No abstract available. PMID 30180376
- [Background] Frantzidis CA, Vivas AB, Tsolaki A, Klados MA, Tsolaki M, Bamidis PD. Functional disorganization of small-world brain networks in mild Alzheimer's Disease and amnestic Mild Cognitive Impairment: an EEG study using Relative Wavelet Entropy (RWE). Front Aging Neurosci. 2014 Aug 26;6:224. doi: 10.3389/fnagi.2014.00224. eCollection 2014. PMID 25206333
- [Background] Konstantinidis EI, Billis AS, Mouzakidis CA, Zilidou VI, Antoniou PE, Bamidis PD. Design, Implementation, and Wide Pilot Deployment of FitForAll: An Easy to use Exergaming Platform Improving Physical Fitness and Life Quality of Senior Citizens. IEEE J Biomed Health Inform. 2016 Jan;20(1):189-200. doi: 10.1109/JBHI.2014.2378814. PMID 26731797
- [Background] Whitfield-Gabrieli S, Thermenos HW, Milanovic S, Tsuang MT, Faraone SV, McCarley RW, Shenton ME, Green AI, Nieto-Castanon A, LaViolette P, Wojcik J, Gabrieli JD, Seidman LJ. Hyperactivity and hyperconnectivity of the default network in schizophrenia and in first-degree relatives of persons with schizophrenia. Proc Natl Acad Sci U S A. 2009 Jan 27;106(4):1279-84. doi: 10.1073/pnas.0809141106. Epub 2009 Jan 21. PMID 19164577
- [Result] Arbabshirani MR, Kiehl KA, Pearlson GD, Calhoun VD. Classification of schizophrenia patients based on resting-state functional network connectivity. Front Neurosci. 2013 Jul 30;7:133. doi: 10.3389/fnins.2013.00133. eCollection 2013. PMID 23966903
- [Result] Bamidis PD, Fissler P, Papageorgiou SG, Zilidou V, Konstantinidis EI, Billis AS, Romanopoulou E, Karagianni M, Beratis I, Tsapanou A, Tsilikopoulou G, Grigoriadou E, Ladas A, Kyrillidou A, Tsolaki A, Frantzidis C, Sidiropoulos E, Siountas A, Matsi S, Papatriantafyllou J, Margioti E, Nika A, Schlee W, Elbert T, Tsolaki M, Vivas AB, Kolassa IT. Gains in cognition through combined cognitive and physical training: the role of training dosage and severity of neurocognitive disorder. Front Aging Neurosci. 2015 Aug 7;7:152. doi: 10.3389/fnagi.2015.00152. eCollection 2015. PMID 26300772
- [Result] Frantzidis CA, Ladas AK, Vivas AB, Tsolaki M, Bamidis PD. Cognitive and physical training for the elderly: evaluating outcome efficacy by means of neurophysiological synchronization. Int J Psychophysiol. 2014 Jul;93(1):1-11. doi: 10.1016/j.ijpsycho.2014.01.007. Epub 2014 Jan 25. PMID 24472698
- [Result] Rosazza C, Minati L. Resting-state brain networks: literature review and clinical applications. Neurol Sci. 2011 Oct;32(5):773-85. doi: 10.1007/s10072-011-0636-y. Epub 2011 Jun 11. PMID 21667095